CLINICAL TRIAL: NCT05314127
Title: Efficacy of Tazarotene Versus Topical 5-Fluorouracil, and Imiquimod in The Treatment of Verruca Plana
Brief Title: Efficacy of Tazarotene in Treatment of Verruca Plana
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hagar Nofal, Lecturer, Principal Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9326/22-2-2022
Record Dates: First submitted 2022-03-20; First posted 2022-04-06 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Warts Flat
MeSH Terms: interventions — tazarotene; Imiquimod; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Tazarotene (Experimental): 20 patients of verruca plana receiving daily topical Tazarotene 0.1% gel at night
  Interventions: Drug: Tazarotene 0.1% Gel,Top
- Imiquimod (Active Comparator): 20 patients with verruca plana will be treated with imiquimod cream 5% applied once daily at night
  Interventions: Drug: Imiquimod
- 5- fluorouracil (Experimental): 20 patients with verruca plana will be treated with topical 5- fluorouracil 5% cream applied once daily at night
  Interventions: Drug: Fluorouracil Cream
- Petrolatum (Placebo Comparator): 20 patients with verruca plana will be treated with petroleum jelly once daily at night.
  Interventions: Drug: Petrolatum

INTERVENTIONS:
Drug: Tazarotene 0.1% Gel,Top — once daily topical application at night with a cotton tipped applicator on every lesion
  Arms: Tazarotene
Drug: Imiquimod — Imiquimod cream 5% applied once daily at night with a cotton tipped applicator applied once daily.
  Arms: Imiquimod
Drug: Fluorouracil Cream — 5- Fluorouracil Cream 5% is applied once daily at night with a cotton tipped applicator
  Arms: 5- fluorouracil
Drug: Petrolatum — applied once daily at night
  Arms: Petrolatum

SUMMARY:
Verruca plana is a common skin infection with worldwide distribution. Approximately 10% of general population is infected with flat warts and it represents up to 18 % of the patients seeking treatment for warts. Verruca plana is not merely an infectious disease but also affects the quality of patients' life. Verruca plana causes major cosmetic and social concerns. Lesions' persistence and recurrence cause frustrations and psychological distress which motivate patients to seek different treatment strategies. Verruca plana commonly affects the school aged children which augments its effect on the psychological and social development of children with stigmatization and bullying are great risks. The available treatment strategies neither ensured complete clearance of the disease nor were free of side effects. Frequently used physical removal methods are operator dependent and commonly lead to irritation, local inflammation, scars, dyspigmentation, and disfigurement. In this study we evaluate the efficacy and the safety of tazarotene gel 0.1% in the treatment of verruca plana compared to imiquimod or 5-fluorouracil

DETAILED DESCRIPTION:
Patients will be assigned randomly into one of 4 groups as 1:1:1:1 using randomization.com with the seed number 7607

* Group (A): Patients will be treated with topical tazarotene gel 0.1%with a cotton tipped applicator on every lesion once daily at night.
* Group (B): Patients will be treated with topical 5- fluorouracil 5% cream applied once daily at night.
* Group (C): Patients will be treated with imiquimod cream 5% applied once daily at night.
* Group (D): Patients will be treated with petroleum jelly once daily at night.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be willing to sign informed consent; for patients younger than 18 years old, parents or guardians will sign an informed consent

  * Age > 4 years.
  * Both sexes.
  * Patients with clinically and dermoscopically diagnosed plane warts.
  * Subject is willing and able to follow all study instructions and to attend all study visits

Exclusion Criteria:

* • History of hypersensitivity to any of the drugs used.

  * Pregnancy and lactation.
  * Patients with epidermodysplasia verruciformis syndrome.
  * Patients with eczematous skin disorders.
  * Presence of any active infections e.g. herpes, tuberculosis.
  * History of topical anti wart treatment within 4 weeks of recruitment to the study, and a 12-week period for systemic anti-wart treatment, or immunotherapy, or HPV vaccine in the last 24 weeks.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with complete clearance of flat warts (Physician Wart Assessment scale PWA = 0) at the end in the four arms of the clinical trial. | Till complete clearance of all lesions or a maximum of 12 weeks, whichever came first
  Complete clearance is defined by complete disappearance of the warts and return to normal skin markings
The incidence of adverse events measured by the percentage of participants developing them in the four arms of the study | Till complete clearance of all lesions or a maximum of 12 weeks, whichever came first

SECONDARY OUTCOMES:
The mean percent of warts achieving PWA 0 (complete clearance) per-participant across the different arms of the clinical trial | Till complete clearance of all lesions or a maximum of 12 weeks, whichever came first
The median time for participants to achieve clearance of all warts in the different arms of the clinical trial. | Till complete clearance of all lesions or a maximum of 12 weeks, whichever came first
The proportion of patients achieving poor response (<50% of warts disappeared) or partial response (> 50%-99% of warts disappeared) | Till complete clearance of all lesions or a maximum of 12 weeks, whichever came first
The quality of life index measured by the difference in the wart specific Dermatology Life Quality Index at the end of the trial compared to the baseline | at the end of 6 months period follow up
The patients' adherence to treatment measured by the percentage of patients withdrawn from each arm of the trial | at the end of 12 weeks study period
The patients' adherence to treatment measured by the percentage of missed doses in each arm of the trials | at the end of 12 weeks study period

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology department, Zagazig University Hospitals, Faculty of Medicine, Zagazig University, Zagazig, Select Region, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Hodeib AAE, Al-Sharkawy BG, Hegab DS, Talaat RAZ. A comparative study of intralesional injection of Candida albicans antigen, bleomycin and 5-fluorouracil for treatment of plane warts. J Dermatolog Treat. 2021 Sep;32(6):663-668. doi: 10.1080/09546634.2019.1688236. Epub 2019 Nov 12. PMID 31682472
- [Background] Gladsjo JA, Alio Saenz AB, Bergman J, Kricorian G, Cunningham BB. 5% 5-Fluorouracil cream for treatment of verruca vulgaris in children. Pediatr Dermatol. 2009 May-Jun;26(3):279-85. doi: 10.1111/j.1525-1470.2008.00800.x. PMID 19706088
- [Background] Kim MB, Ko HC, Jang HS, Oh CK, Kwon KS. Treatment of flat warts with 5% imiquimod cream. J Eur Acad Dermatol Venereol. 2006 Nov;20(10):1349-50. doi: 10.1111/j.1468-3083.2006.01709.x. No abstract available. PMID 17062069
- [Background] Nofal A, Marei A, Ibrahim AM, Nofal E, Nabil M. Intralesional versus intramuscular bivalent human papillomavirus vaccine in the treatment of recalcitrant common warts. J Am Acad Dermatol. 2020 Jan;82(1):94-100. doi: 10.1016/j.jaad.2019.07.070. Epub 2019 Jul 29. PMID 31369771